CLINICAL TRIAL: NCT02967315
Title: Effects of Changes in Fluid Status on Right Ventricular Volumes and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-0399; 2013-0276 (Other: HS IRB); SMPH/SURGERY/CARDIOTHORACIC (Other: A539782)
Record Dates: First submitted 2016-10-27; First posted 2016-11-18 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot | interventions — X-Rays; Hypodermoclysis; Blood Specimen Collection; Pregnancy Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Procedures include:
  Two Cardiac Magnetic Resonance Imaging (CMRIs) A central venous line placement, A chest X-ray Electrocardiogram (ECG) Fluid administration Blood draw Pregnancy test
  Interventions: Procedure: Cardiac Magnetic Resonance Imaging (CMRI); Procedure: Central venous line placement; Procedure: Chest X-ray; Procedure: Fluid administration; Procedure: Blood Draw; Procedure: Pregnancy test; Procedure: Electrocardiogram

INTERVENTIONS:
Procedure: Cardiac Magnetic Resonance Imaging (CMRI) — There will be 2 CMRIs. The first one will be patient's routine clinically schedule CMRI after the patient has fasted for 12 hours.This CMRI uses contrast.
  The second CMRI will be the research CMRI after the fluid administration. This CMRI does not use contrast.
Procedure: Central venous line placement — An ultrasound guided central line catheter will be placed in the internal jugular vein (IJV) under local anesthesia.
Procedure: Chest X-ray — A chest X-ray will be performed for safety reasons to rule out pneumothorax (< 1% risk) after central line placement.
Procedure: Fluid administration — Administration of 15cc/kg of normal saline for fluid hydration through peripheral IV that is placed for the MRI contrast administration.
Procedure: Blood Draw — One to two teaspoons of blood will be drawn for basic metabolic panel.
Procedure: Pregnancy test — A urine pregnancy test will be performed in female subjects.
Procedure: Electrocardiogram — 12 lead ECG

SUMMARY:
The purpose of this study is to evaluate the correlation between fluid volume status and right ventricular volume and function, in those with free pulmonary valve insufficiency after Tetralogy of Fallot (TOF) repair.

DETAILED DESCRIPTION:
The purpose of this study is to measure the changes in Right Ventricular size and function with changes in preload, using cardiovascular magnetic resonance (CMR). Based on an intensive research and clinical observations the investigators hypothesize that changes in volume status cause a statistically significant difference in the Cardiovascular magnetic resonance (CMR) measured RV End Diastolic Volume (EDV), end-systolic volume (ESV), ejection fraction (EF) and pulmonary regurgitation (PR). The investigator hypothesizes that smaller changes will occur in left ventricular LV EDV, ESV, and EF.

1. To establish a correlation between the changes in preload volume status and RV size and function in patients with free pulmonary insufficiency (PI) after TOF repair using CMRI.
2. To assess the effects of preload status on the measured severity of pulmonary regurgitation (PR).
3. To assess the effects of preload status on the left ventricular (LV) size

This study will be conducted in compliance with this protocol, good clinical practice and the applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. TOF patients who have had repair using a transannular patch.
2. Patients that present with free pulmonary insufficiency.
3. Are older than 18 years.

Exclusion Criteria:

1. Patients who have lesions predisposing to chronic volume overload (i.e. patients with significant residual postoperative ventricular septal defects (VSD), or large aorto-pulmonary collaterals or more than moderate tricuspid insufficiency) since all these hemodynamic conditions can influence the late function of the right ventricle and potentially affect the response of the right side of the heart in changes in volume status
2. Patients who had a valve sparing TOF repair and have less than free pulmonary insufficiency.
3. Patients who have significant residual right-sided obstruction (i.e. patients who have residual RVOT obstruction or significant residual branch pulmonary artery stenosis), as it is shown that residual pulmonary stenosis may protect from RV dilation and from deterioration of the RV function.
4. Patients who cannot be reconstructed with a transannular patch and/or require a right ventricle to pulmonary artery homograft for reconstruction including:

   * pulmonary atresia and VSD
   * patients with anomalous coronary crossing the right ventricular outflow tract (RVOT) and
   * patients with TOF-absent pulmonary valve syndrome.
5. Patients with renal failure and renal insufficiency
6. Patients with uncompensated heart failure
7. Cancer patients
8. Latex allergic patients
9. Patients with diabetes
10. Pregnant females
11. Prisoners
12. Individuals who lack consent capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Postload volume status | 24 months
  The following will be measured to define the postload volume status: Left and right ventricle end diastolic volume (milliliters [ml]); Ejection fraction (%); pulmonary regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: Petros V Anagnostopoulos, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No